CLINICAL TRIAL: NCT02016222
Title: Tear Analysis in the Diagnosis of Primary Progressive Forms of Multiple Sclerosis
Brief Title: Tear Analysis in the Diagnosis of Multiple Sclerosis
Acronym: LARMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0006
Record Dates: First submitted 2013-11-22; First posted 2013-12-19 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Primary Progressive Multiple Sclerosis
Keywords: primary progressive multiple sclerosis; diagnosis; tears; isoelectric focusing; oligoclonal bands
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Disease; Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tears sampling (Experimental)
  Interventions: Procedure: tears sampling

INTERVENTIONS:
Procedure: tears sampling

SUMMARY:
In the primary progressive multiple sclerosis, the detection of oligoclonal bands in cerebrospinal fluid is critical for the diagnosis. However, lumbar puncture for cerebrospinal fluid collection is considered relatively invasive. Our hypothesis is that oligoclonal bands detection in tears is possible and useful for the diagnosis of multiple sclerosis.

DETAILED DESCRIPTION:
The objective of the present study is to assess concordance between oligoclonal bands detection in tears and in cerebrospinal fluid. We will include patients with primary progressive multiple sclerosis and we will compare results of oligoclonal bands detection by isoelectric focusing in cerebrospinal fluid and tears. Tears will be collected using a Schirmer strip. This would circumvent the practice of invasive lumbar punctures currently used in multiple sclerosis diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Progressive neurological deficit after 12 months
* At least 9 T2 brain lesions of minimum 3 mm evidenced by MRI and/or four or more T2 lesions of minimum 3 mm with positive Visual Evoked Potential and/or positive spinal cord MRI (at least two focal T2 lesions)

Exclusion Criteria:

* Asiatic persons
* recurrent forms of the disease
* Persons wearing contact lenses
* Ocular Infection
* Corticoid treatment at least 30 days before sampling
* immunosuppressive or immunomodulatory treatment 3 months before sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Concordance between the quantification of oligoclonal IgG bands by isoelectric focusing in tears and in the cerebrospinal fluid in patients with primary progressive multiple sclerosis | at baseline and two years after (+/- 2 months)

SECONDARY OUTCOMES:
Isoelectrophoretic profile of tears | Baseline and two years after inclusion
  Determination of the stability and prognostic value of isoelectrophoretic profile of tears at inclusion, after 2 years.
Isoelectrophoretic profiles of tears by digital recording and analysis of images | Baseline and two years after

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hautecoeur, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille (GHICL); Elisabeth Baumelou, MD, Study Chair — Groupement des Hôpitaux de l'Institut Catholique de Lille; Patrick Vermersch, MD, PhD, Principal Investigator — Centre Hospitalier Régional, Universitaire de Lille; Christine Lebrun-Frenay, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice; Jérome De Sèze, MD, PhD, Principal Investigator — Centre Hospitalier Régional Universitaire de Strasbourg; Thibaut Moreau, MD, Principal Investigator — Centre Hospitalier Universitaire Dijon; Pierre Clavelou, MD, Principal Investigator — Centre Hospitalier Régional Universitaire de Clermont-Ferrand; Olivier Heinzlef, MD, Principal Investigator — Centre hospitalier intercommunal de Poissy; Christian Confavreux, MD, Principal Investigator — Hospices Civils de Lyon; Marc Debouverie, MD, PhD, Principal Investigator — Central Hospital, Nancy, France; Jean Pelletier, MD, PhD, Principal Investigator — L'assistance Publique des Hôpitaux de Marseille; Bruno Brochet, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Gilles Defer, MD, Principal Investigator — Centre Hospitalier Universitaire de Caen; Eric Thouvenot, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (13):
- France (13):
  - Centre hospitalier universitaire (CHU), Nice, Nice, Alpes Maritimes
  - Groupement des Hôpitaux de l'Institut Catholique de Lille (GHICL), Lille, Nord
  - Centre hospitaliere universitaire, Bordeaux
  - Centre hospitalier universitaire, Caen
  - Centre hospitalier régional universitaire, Clermont-Ferrand
  - Centre hospitalier universitaire, Dijon
  - Centre hospitalier régional universitaire, Lille
  - Hospices civils de Lyon, Lyon
  - Assistance Publique - Hôpitaux de Marseille, Marseille
  - Centre hospitalier universitaire, Nancy
  - Centre hospitalier universitaire, Nîmes
  - Centre hospitalier intercommunal, Poissy
  - Centre hospitalier régional universtaire, Strasbourg